CLINICAL TRIAL: NCT00044642
Title: Long-Term Lorazepam Use and Acute Toxicity in the Aged
Brief Title: Lorazepam-Induced Toxicity in the Aged
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: R01MH059142 (NIH); R01MH059142 (NIH); DATR A4-GPX
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Anxiety Disorders; Generalized Anxiety Disorder
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Lorazepam

INTERVENTIONS:
Drug: Lorazepam

SUMMARY:
This study will compare the effects of an acute dose of lorazepam to a placebo in elderly patients with generalized anxiety disorder (GAD).

DETAILED DESCRIPTION:
GAD is among the most common anxiety disorders in the elderly population. The drug lorazepam is widely utilized in the treatment of elderly individuals with GAD. However, single doses of lorazepam have been associated with cognitive toxicity that is typically evident between 1 and 2.5 hours after the drug is administered. The toxic effects include decreased memory and increased swaying, which has been associated with greater risk for falls.

Patients have 4 study visits. A psychiatric evaluation and a memory test are given at the first visit. During the second study visit, patients have a physical exam, an electrocardiogram (ECG), a neuropsychological assessment, an optional magnetic resonance imaging (MRI) brain scan, and other laboratory tests. On the third and fourth visits, patients are randomized to receive either their highest daily dose of lorazepam or placebo. Performance effects and postural sway are determined before drug administration and at 1, 2.5, and 5 hours after the drug is given. Blood samples for the determination of drug levels are also obtained.

ELIGIBILITY:
Inclusion Criteria:

* Lorazepam treatment for at least 3 months
* Cognitively intact

Note: Individuals who are unable or unwilling to have an MRI may be included

Exclusion Criteria:

* Major psychiatric disorder other than GAD
* Significant medical illness which may increase the likelihood of adverse reactions to lorazepam
* Severe loss of hearing or vision
* Current or past history of alcohol dependence
* Substance abuse within the past 6 months
* MRI evidence of infection, infarction, or other lesions suggestive of intervening neurological disease
* Clinical symptoms that suggest neurological disease
* Dementia or other mental syndromes or disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2000-12; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nunzio Pomara, MD, Principal Investigator — Nathan S. Kline Institute and New York University School of Medicine
Locations (2):
- United States (2):
  - NYU/Bellevue General Clinical Research Center (8East), New York, New York
  - Nathan S. Kline Institute, Orangeburg, New York

REFERENCES:
- See also: Nathan S. Kline Institute for Psychiatric Research — http://www.rfmh.org/nki/